CLINICAL TRIAL: NCT07357454
Title: Evaluation of the Smart Talk: Cannabis Awareness and Prevention Curriculum
Brief Title: Smart Talk: Cannabis Awareness and Prevention Curriculum Evaluation
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Bonnie Halpern-Felsher, Professor of Pediatrics, Stanford School of Medicine, Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 80402; 1R01DA060900-01A1 (NIH)
Record Dates: First submitted 2026-01-20; First posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2025-11

CONDITIONS: Cannabis Use
Keywords: youth cannabis education health prevention

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Smart Talk Cannabis Awareness and Prevention (Experimental): At the start of Year 2, schools will be randomized in a 1:1 ratio to either receive 'Stanford REACH Lab's Smart Talk: Cannabis Prevention and Awareness' curriculum or 'delay-in-treatment (standard of care)'. Students in these schools will receive the Stanford curriculum designed as a 5-session course administered in a school class-room setting.
  Interventions: Behavioral: Behavioral: Smart Talk Cannabis Awareness and Prevention
- Delay in Treatment Group (Experimental): At the start of Year 2, schools randomized to the delay-in-treatment group will receive a standard of care for one year. After year 2, the delay-in-treatment group will crossover to receive 'Stanford REACH Lab's Healthy Futures: Cannabis Prevention and Awareness until year 5 (receive intervention for years 2 to 4).
  Interventions: Behavioral: Behavioral: Smart Talk Cannabis Awareness and Prevention

INTERVENTIONS:
Behavioral: Behavioral: Smart Talk Cannabis Awareness and Prevention — Behavioral:Smart Talk includes 5 lessons, each providing activities, online quiz games, and worksheets in addition to presentations, resources, and other materials aimed at addressing key factors associated with youth cannabis use, including changing adolescents' attitudes towards and misperceptions about cannabis; increasing their refusal skills to pulls of marketing and social media; reducing stress and depression which have been linked to cannabis initiation and use; improving coping skills; and decreasing intentions and actual use of all cannabis products.

SUMMARY:
The Stanford REACH Lab's SMART TALK: Cannabis Awareness and Prevention Toolkit is a free, online educational resource to be used by educators to increase knowledge and awareness of cannabis and reduce use among youth. The aim of this study is to investigate the extent to which the curriculum changes middle and high school students' intentions to use and actual use of cannabis.

DETAILED DESCRIPTION:
Smart Talk includes 5 lessons, each providing activities, online quiz games, and worksheets in addition to presentations, resources, and other materials aimed at addressing key factors associated with youth cannabis use, including changing adolescents' attitudes towards and misperceptions about cannabis; increasing their refusal skills to pulls of marketing and social media; reducing stress and depression which have been linked to cannabis initiation and use; improving coping skills; and decreasing intentions and actual use of all cannabis products.

ELIGIBILITY:
Inclusion Criteria:

* Middle school and high school students receiving health education at schools participating in the study

Exclusion Criteria:

-

Ages: 10 Years to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 10800 (Estimated)
Dates: Start 2026-08 (Estimated); Primary Completion 2029-09 (Estimated); Study Completion 2030-02 (Estimated)

PRIMARY OUTCOMES:
Change in cannabis use | Baseline to follow-up at approximately 182 weeks
  Investigator-originated survey measures (questions) assess ever cannabis use & past 30-day cannabis use. This outcome measure assesses cannabis use.

SECONDARY OUTCOMES:
Change in intention to use cannabis in the future | Baseline to follow-up at approximately 182 weeks
  Investigator-originated survey measures (questions) assessing change in participant intention to use cannabis in the future

CONTACTS AND LOCATIONS:
Overall Officials: Bonnie Halpern Felsher, Ph.D., Principal Investigator — Stanford University
Locations (1):
- Stanford University, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No